CLINICAL TRIAL: NCT03621514
Title: The Feasibility and Advantages of Painless Indwelling Catheter in Uniportal Video-assisted Thoracoscopic Surgery Lobectomy of Lung Cancer: A Prospective Cohort Study
Brief Title: The Feasibility and Advantages of Painless Indwelling Catheter in Uniportal VATS Lobectomy of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xueying Yang (Other)
Responsible Party: Sponsor-Investigator, Xueying Yang, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2018-KS-032
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Urethral Catheter; Complications
Keywords: Painless indwelling urethral catheter; uniportal video-assisted thoracoscopic surgery; Lobectomy; Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Catheters, Indwelling

STUDY DESIGN:
Intervention Model Description: This study is a prospective cohort study.The main study content is the feasibility and advantages of painless indwelling catheter in perioperative period of uniportal video-assisted thoracoscopic surgery in lobectomy of lung cancer,divided into exposed and non-exposed groups.The exposed group was painless indwelled urethral catheter, the non-exposed group was indwelled urethral catheter routinely.
Who Masked: Outcomes Assessor
Masking Description: This study is a prospective cohort study.Participants,Care Provider, and Investigator all know the grouping situation. The Investigator collect the information and observation indicators of the two groups of participants and send to the Outcomes Assessor . The Outcomes Assessor does not know the grouping situation of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- painless indwelling catheter (Other): This group of patients underwent catheterization after anesthesia. At the end of the operation, the patient was removed from the catheter before anesthesia was awakened.
  Interventions: Procedure: painless indwelling catheter
- indwelling catheter (Other): This group of patients underwent catheterization after anesthesia,and the catheter was indwelled. The patient was routinely removed for 24 to 72 hours after surgery.
  Interventions: Procedure: indwelling catheter

INTERVENTIONS:
Procedure: painless indwelling catheter — Catheterization after anesthesia (14 F Foley's urinary catheter), the patient was removed before the anesthesia was awakened and the catheter was removed(Fully lubricate the anterior end of the catheter with a lidocaine ointment 2.5g before catheterization).
  Other Names: 14 F Foley's catheter; lidocaine ointment
  Arms: painless indwelling catheter
Procedure: indwelling catheter — The patients underwent catheterization(14 F Foley's catheter) after anesthesia,and the catheter was indwelled(Fully lubricate the anterior end of the catheter with a lidocaine ointment 2.5g before catheterization). The patient was routinely removed for 24 to 72 hours after surgery.
  Other Names: 14 F Foley's catheter; lidocaine ointment
  Arms: indwelling catheter

SUMMARY:
This study is a prospective cohort study.The main study content is the feasibility and advantages of painless indwelling catheter in perioperative period of uniportal video-assisted thoracoscopic surgery in lobectomy of lung cancer,divided into exposed and non-exposed groups.The exposed group was painless indwelled urethral catheter, the non-exposed group was indwelled urethral catheter routinely.

DETAILED DESCRIPTION:
This study is a prospective cohort study.The main study content is the feasibility and advantages of painless indwelling catheter in perioperative period of uniportal video-assisted thoracoscopic surgery in radical resection of lung cancer,divided into exposed and non-exposed groups,divided into exposed and non-exposed groups.Communicating with the surgeon and patients who meet the inclusion criteria, decide whether to enter the exposed or non-exposed group.The exposed group was painless indwelled urethral catheter, the non-exposed group was indwelled urethral catheter routinely.By collecting personal information of two groups of patients and the corresponding observation indicators to analyze whether the painless indwelling urethral catheters in lobectomy of lung cancer is more beneficial than the indwelled urethral catheter routinely in lobectomy of lung cancer, and it is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75-year old patient with lung cancer who is eligible for Uniportal Video-assisted Thoracoscopic Surgery in lobectomy.

2.The result of rapid pathology is primary lung cancer.

3.Electrocardiogram, pulmonary function, color Doppler echocardiography, arteriovenous color Doppler ultrasound and other preoperative examination results are normal.

4.The patient agreed to participate in the study and signed the informed consent form.

Exclusion Criteria:

1. Patients have severe urinary system diseases (medium-to-severe BPH, urethral stricture, urinary calculi, infections, tumors, etc.) ,and/or have undergone abdominal and pelvic surgery before surgery.
2. There is a potential infection before surgery.
3. Heart and lung serious organic diseases.
4. Combined thoracic adhesions, patients with severe coagulation insufficiency.
5. The time of anesthesia is more than 4 hours.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Urine retention rate | 10 days
  Urine retention rate

SECONDARY OUTCOMES:
Urinary tract infection | 10 days
  The two groups of patients were each examined for middle urine after extubation. Refer to the clinical diagnostic criteria of the 2006 Hospital Infection Diagnostic Criteria (Trial): If the urinary leukocyte male ≥ 5 / high power field, female ≥ 10 / high power field, accompanied or not accompanied by urinary frequency, urgency, dysuria, etc. Symptoms of urinary tract irritation; or pain in the lower abdomen, pain in the kidney area, with or without fever.
Postoperative bedtime | 2 days
  The time from the patient's postoperative pushback to the first bedtime
Postoperative hospital stay | 15 days
  Postoperative hospital stay
The total cost of hospitalization | 15 days
  The total cost of hospitalization
Postoperative pain level | 3 days
  Using visual analogue scale/score (VAS), the degree of discomfort (pain and urinary sensation) is represented by 11 numbers from 0 to 10, with 0 being painless and no urine, and 10 being the most painful. (or) The sense of urinary sensation is strong, so that the patient can choose the number according to the feeling of self, indicating the degree. 0 degree: 0 points, no discomfort; I degree (mild): 1 to 3 points, with slight pain and/or urinary sensation, can tolerate; II degree (moderate): 4 to 7 points, patient pain And/or urinary sensation and affect sleep, can tolerate; III degree (severe): 8 to 10 points, the patient has progressively strong pain and/or urinary sensation, pain is unbearable, affecting appetite, affecting sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] Caronia FP, Loizzi D, Nicolosi T, Castorina S, Fiorelli A. Tubeless tracheal resection and reconstruction for management of benign stenosis. Head Neck. 2017 Dec;39(12):E114-E117. doi: 10.1002/hed.24942. Epub 2017 Sep 27. PMID 28960733
- [Result] Zhao ZR, Lau RWH, Ng CSH. Anaesthesiology for uniportal VATS: double lumen, single lumen and tubeless. J Vis Surg. 2017 Aug 21;3:108. doi: 10.21037/jovs.2017.07.05. eCollection 2017. PMID 29078668
- [Result] Xia Z, Qiao K, He J. Recent advances in the management of pulmonary tuberculoma with focus on the use of tubeless video-assisted thoracoscopic surgery. J Thorac Dis. 2017 Sep;9(9):3307-3312. doi: 10.21037/jtd.2017.08.44. PMID 29221316
- [Result] Boisen ML, Rao VK, Kolarczyk L, Hayanga HK, Gelzinis TA. The Year in Thoracic Anesthesia: Selected Highlights from 2016. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):791-799. doi: 10.1053/j.jvca.2017.02.182. Epub 2017 Feb 22. No abstract available. PMID 28689818
- [Result] Yang SM, Wang ML, Hung MH, Hsu HH, Cheng YJ, Chen JS. Tubeless Uniportal Thoracoscopic Wedge Resection for Peripheral Lung Nodules. Ann Thorac Surg. 2017 Feb;103(2):462-468. doi: 10.1016/j.athoracsur.2016.09.006. Epub 2016 Nov 16. PMID 27865474
- [Result] Mineo TC, Tamburrini A, Perroni G, Ambrogi V. 1000 cases of tubeless video-assisted thoracic surgery at the Rome Tor Vergata University. Future Oncol. 2016 Dec;12(23s):13-18. doi: 10.2217/fon-2016-0348. Epub 2016 Sep 30. PMID 27686131
- [Result] Gonzalez-Rivas D, Yang Y, Guido W, Jiang G. Non-intubated (tubeless) uniportal video-assisted thoracoscopic lobectomy. Ann Cardiothorac Surg. 2016 Mar;5(2):151-3. doi: 10.21037/acs.2016.03.02. No abstract available. PMID 27134844
- [Result] Peng G, Liu M, Luo Q, Chen H, Yin W, Wang W, Huang J, Qiu Y, Guo Z, Liang L, Dong Q, Xu X, He J. Spontaneous ventilation anesthesia combined with uniportal and tubeless thoracoscopic lung biopsy in selected patients with interstitial lung diseases. J Thorac Dis. 2017 Nov;9(11):4494-4501. doi: 10.21037/jtd.2017.10.76. PMID 29268519
- [Result] Feneley RC, Hopley IB, Wells PN. Urinary catheters: history, current status, adverse events and research agenda. J Med Eng Technol. 2015;39(8):459-70. doi: 10.3109/03091902.2015.1085600. Epub 2015 Sep 18. PMID 26383168
- [Result] Petersen RH, Holbek BL, Hansen HJ, Kehlet H. Video-assisted thoracoscopic surgery-taking a step into the future. Eur J Cardiothorac Surg. 2017 Apr 1;51(4):694-695. doi: 10.1093/ejcts/ezw381. No abstract available. PMID 28007878
- [Result] Tobu S, Noguchi M, Hashikawa T, Uozumi J. Risk factors of postoperative urinary retention after hip surgery for femoral neck fracture in elderly women. Geriatr Gerontol Int. 2014 Jul;14(3):636-9. doi: 10.1111/ggi.12150. Epub 2013 Nov 12. PMID 24215579
- [Result] Assadi F. Strategies for Preventing Catheter-associated Urinary Tract Infections. Int J Prev Med. 2018 Jun 4;9:50. doi: 10.4103/ijpvm.IJPVM_299_17. eCollection 2018. No abstract available. PMID 29963301
- [Derived] Zhang L, Yang X, Tian Y, Yu Q, Xu Y, Zhou D, Wu Z, Zhao X. The feasibility and advantages of immediate removal of urinary catheter after lobectomy: A prospective randomized trial. Nurs Open. 2021 Nov;8(6):2942-2948. doi: 10.1002/nop2.1006. Epub 2021 Jul 30. PMID 34329541